CLINICAL TRIAL: NCT06744049
Title: Assessment of Transfer Direct System (TDS) as a New Method for Embryo Transfer
Brief Title: Transfer Direct System as a New Method for Embryo Transfer
Acronym: TDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Premium Fertility (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PF-TDS-XS-23-01
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Embryo Transfer
Keywords: Semi-automatization; Embryo implantation

STUDY DESIGN:
Intervention Model Description: Clinical research with medical device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Embryo transfer with Transfer Direct System (TDS) (Experimental): The trial has a single assignment group aimed at patients of reproductive age who attend the clinic with a desire for a child and undergo Assisted Reproduction Treatment (ART) with an euploid single embryo transfer (SET) after corresponding hormone replacement therapy (HRT) has been carried out.
  Interventions: Device: Transfer Direct System (TDS)

INTERVENTIONS:
Device: Transfer Direct System (TDS) — Class IIA medical device (according to rule 5 of Annex VIII of Regulation (EU) 2017/745 for medical devices). A semi-automated medical equipment designed to inject an embryo into the maternal uterine endometrium through the lumen of the female reproductive system.

SUMMARY:
Infertility is defined as the inability to conceive within a year of unprotected intercourse. Infertility affects one in six couples and represents a public health problem causing feelings of helplessness, depression, and anxiety in both women and men worldwide. Despite the desire to become parents, up to 50% of infertile couples do not seek medical treatment, and 50-60% abandon treatment after two or three failed in vitro fertilization (IVF) cycles, even when the procedure is covered by insurance or public health. There are multiple reasons for this discontinuation; however, after removing cost considerations, psychological stress and poor prognoses represent the main reasons for stopping treatment.

Clinical infertility treatments are generally ineffective. Success remains poor even with IVF, as evidenced by current live birth rates (LBRs) of only ~30% per initiated cycle. The primary challenge in ART lies mainly in the embryo implantation process, which remains the most significant bottleneck in IVF success, accounting for over 50% of ART failures.

Embryo transfer (ET), the final step in IVF, has seen little technological advancement since its inception over four decades ago. The procedure is typically performed transcervically and largely relies in tactile sensation and operator's experience. Although a simple procedure, several potential negative factors may be linked to the low number of IVF pregnancies, including variations in catheter placement, the risk of uterine contractions and lack of control of intrauterine pressure and embryo placement can result in up to 15% of the transferred embryos being inadvertently expelled from the uterus. Therfore, ET's success is highly dependent on non-controllable variables as well as the skill and experience of the operator, resulting in significant inter-operator variability.

Premium Fertility team has developed a controlled embryo transfer system - the Transfer Direct System (TDS) - that incorporates a visualization system to guide embryo delivery with the help of a fully automated microfluidic system that avoids initial phases of apposition and adhesion of implantation of human embryos. This technique places the embryo directly in the endometrial tissue, thereby minimizing the effects of embryo expulsion and potentially offering significant advantages such as the ability to visualize the uterine cavity through an endoscope at the time of embryo transfer and control the mechanics of the injection procedure to increase precision.

DETAILED DESCRIPTION:
Embryo transfer represents the most critical step in IVF; however, this highly operator-dependent procedure has not evolved significantly since the first description of its use. In this study, Premium Fertility investigators propose a new method of embryo transfer using high-precision automated injection of embryos into the uterus to minimize expulsion, facilitate implantation, and minimize inter- and intra-operator variability. If successful, TDS will provide for safe and consistent embryo transfer and will be transformative in the most critical procedure of fertility treatments, potentially increasing the success rates of such therapies.

The TDS is a medical device used in embryo transfer processes in patients undergoing ART, and it's a semi-automated piece of medical equipment designed to inject an embryo or a fertilized ovum into the maternal uterine endometrium through the lumen of the female reproductive system. The system is made up of two instruments and different consumables:

* CEC device: an instrument embryologists use to collect the human embryo for transfer and performs the functions of wetting the needle and collecting the embryo. This instrument does not interact with the patient.
* CET device: an instrument gynecologists use to inject an embryo into the maternal uterine endometrium. This instrument is placed in the embryo transfer room and has an umbilical cable controlling the TD needle that ultimately injects the embryo in the endometrial tissue. None of the CET components come into direct or indirect contact with the patient.
* Consumables:

  * TD needle: Performs embryo collection in the embryology laboratory and embryo injection into the maternal uterine endometrium.
  * TD catheter: Used to introduce the TD needle and TD camera through the lumen of the female reproductive system during the transfer; the TD catheter is fixed using the TD speculum lock to keep the needle in stable position during the automatic injection of the embryo. It has a membrane tip at the distal end.
  * TD speculum lock: Fixing the TD catheter to the speculum allows TD catheter placement; manual blocking when it contacts the endometrium ensures a fixed position of the catheter and needle for embryo injection.
  * TD camera: Video and lighting using fiber optics improve the visibility of the vaginal mucosa and the location of the endometrium surface for correct implantation.

The aim of the study is to assess whether the medical device - Transfer Direct System (TDS) - is a safe and effective method for embryo transfer.

This is a prospective, open-label, controlled, non-randomized, multi-center, intervention clinical trial with a Class IIA medical device. The trial has a single assignment group aimed at patients of reproductive age who attend the clinic with a desire for a child and undergo Assisted Reproduction Treatment (ART) with an euploid single embryo transfer (SET) after corresponding hormone replacement therapy (HRT) has been carried out. The inclusion of 80 patients in the study group is expected and will be recruited in at least 2 reference IVF clinics.

Anonymized data from patients receiving euploid single embryo transfer will be used as a control group. For this purpose, data of patients that accomplished the same inclusion criteria will be analysed.

The total expected duration of the study is estimated to be approximately 12 months:

* Six months of recruitment period.
* Three months of approximate total duration of the treatment for each patient.
* Four months to analyze the results, make conclusions, and prepare the final report (overlapped with previous phase).

The study consists of 5 visits:

V1. Starting visit: the Informed Consent Form will be obtained for those patients who come to the clinic to undergo Assisted Reproduction Treatment with Single Embryo Transfer and meet the selection criteria.

V2. Ultrasound and blood test monitoring: the patients will undergo endometrial preparation according to usual clinical practice, preferably with HRT.

V3. Transfer visit: during this visit, embryo transfer will be performed with TDS. Next, the patient will be specifically asked to assess the degree of pain or discomfort from the procedure using an EVA chart, and uterine contractions will be assessed with ultrasound before and after embryo transfer.

V4. Beta performance visit: once the embryo transfer is complete, β-hCG levels will be measured on a blood sample between 10 and 12 days after transfer.

V5. Final visit: in the event of an ongoing pregnancy, a gestational control will be carried out between weeks 8-10 of gestation.

Data will be registered in an electronic Case Report Form (eCRF) specifically designed for this study. Monitoring activities and data verification will be performed during the whole study to ensure data quality, integrity and transparency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose written informed consent is obtained, approved by the Ethics Committees for Investigation with Medicinal Products (ECRmp) after being duly informed of the nature of their disease and after voluntarily accepting the treatment program, knowing the potential risks, benefits, and inconveniences.
2. Patients who are going to undergo ART with a SET and have at least one vitrified euploid blastocyst with PGT-A (Preimplantation Genetic Test for the detection of Aneuploidy).
3. Women of reproductive age between 18 and 50 years (both inclusive)
4. Body mass index (BMI): <30 kg/m2
5. Absence of adenomyosis and endometriosis
6. Uterus without pathologies that can contraindicate the transfer or may hinder implantation (e.g., polyps, fibroids that come into contact with the cavity, or Asherman syndrome) or without a history of thin endometrium or irregular patterns in thin endometrial preparations.
7. Absence of immune pathologies (e.g., lupus) that could endanger the health of the patient.
8. Easy transfer test or history of embryo transfer without difficulty or factors that indicate that the transfer is easy.

Exclusion Criteria:

1. Difficult or very painful transfer tests.
2. Pathologies of an oncological nature.
3. The existence of serious or uncontrolled bacterial, fungal, or viral infections that, in the opinion of the principal investigator, may interfere with the patient's participation in the study or the evaluation of its results.
4. Other circumstances or difficulties that, in the opinion of the investigator, may pose a risk to the subject or reduce the chances of obtaining satisfactory data to achieve the objectives of the study, such as a history of severe preeclampsia without assessment by the obstetric team, psychiatric pathologies without prior assessment by the psychiatrist, uncontrolled or destabilized cardiac pathologies.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients from 18 to 50 years of age without any disease that will undergo ART.
Enrollment: 80 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Safety of TDS in comparison with conventional transfer | From enrollment to final study visit at 8-10 weeks of pregnancy
  Incidence, prevalence and frequency of adverse events.

SECONDARY OUTCOMES:
Efficacy and non-inferiority of TDS | up to 8-10 weeks
  Implantation rate
pregnancy rate | From enrollment to final study visit at 8-10 weeks of pregnancy
  Efficacy and non-inferiority of TDS
ongoing gestation rate | From enrollment to final study visit at 8-10 weeks of pregnancy
  Efficacy and non-inferiority of TDS
miscarriage rate | From enrollment to final study visit at 8-10 weeks of pregnancy
  Efficacy and non-inferiority of TDS

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Eugin Barcelona, Barcelona
  - Clínica Vida Recoletas Sevilla, Seville
  - Clínica Next Fertility Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No